CLINICAL TRIAL: NCT02380989
Title: Integrative Ayurveda Healing Relieves Minor Sports Injury Pain:Results of a Multicenter Controlled Clinical Trial
Brief Title: Integrative Ayurveda Healing Relieves Minor Sports Injury Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adwin Life Care (Industry)
Collaborators: NMP Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Adwin021
Record Dates: First submitted 2015-03-01; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Acute Pain; Sports Injury
Keywords: Ayurveda; Acute pain; Sports Injury
MeSH Terms: conditions — Acute Pain; Athletic Injuries | interventions — Medicine, Ayurvedic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ayurveda (Experimental)
  Interventions: Device: Ayurveda
- Placebo (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Ayurveda — Ayurveda combinations in the form of gel and patches were applied on acute pain site.
  Arms: Ayurveda
Device: Placebo
  Arms: Placebo

SUMMARY:
Sports-related soft tissue injuries, such as sprains, strains, and contusions, are a common painful condition. Current treatment includes oral nonsteroidal anti-inflammatory drugs (NSAIDs), which have a high incidence of intolerable gastrointestinal side effects.

Ancient Indian healing system, Ayurveda addresses the need of sports medicine up to certain extent. In practice, there are different treatment modalities for injuries, uses of drugs & dietetics as well as practices of rehabilitation. Although, previous evidences support the efficacy of ayurveda practices with significant reduction in pain, joint tenderness, joint swelling, mobility restriction and early morning joint stiffness. But there is no treatment studies have been performed to evaluate the clinical outcome for specific sports injuries.

This study assessed the efficacy and safety of ayurveda gel and patches applied to the painful injury site for the treatment of acute minor sports injury pain.

ELIGIBILITY:
Inclusion Criteria:

* inversion ankle injury;
* injury sustained during sporting activity

Exclusion Criteria:

* other lower limb injury;
* concurrent fracture with or without dislocation or with or without complete rupture;
* surgery for ankle injury.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Pain intensity (VAS) | baseline to 3, 7 and 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Archanaben Nachiket, MA, Principal Investigator — NMP Medical Research Institute; Neha Sharma, PhD, Study Director — NMP Medical Research Institute
Locations (3):
- India (3):
  - NMP Medical Research Institute, Mahesāna, Gujarat
  - Khatri educational trust, Satnāli, Haryana
  - GyanSanjeevani, Jaipur, Rajasthan